CLINICAL TRIAL: NCT03814707
Title: Clinical Comparison of Platelet Rich Fibrin Versus Topical Application of Hyaluronic-Acid Gel in Management of Pain And Wound Healing After Free Gingival Graft Harvesting: A Randomized Clinical Trial
Brief Title: Platelet Rich Fibrin VS Hyaloronic Acid in Management of Pain After Harvesting a Free Gingival Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: mostafa soliman (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, mostafa soliman, Principle Investigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-09-17
Record Dates: First submitted 2019-01-13; First posted 2019-01-24 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Pain, Postoperative
Keywords: gingival recession; gingival augmentation; free gingival graft; platelet rich fibrin in wound healing; 2 steps free gingival graft; hyaluronic acid in wound healing
MeSH Terms: conditions — Pain, Postoperative; Gingival Recession

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
  * A randomized clinical trial.
  * Parallel group study.
  * A trial will be carried out in department of periodontology - Faculty of Oral and Dental medicine - Cairo University .
  * Equal randomization : participants with equal probabilities for intervention.
  * Positive controlled : Both groups receiving treatment.
Who Masked: Outcomes Assessor
Masking Description: both the participants and the investigator can't be blinded only outcome assessor will be blinded .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical application 0.2%Hyaluronic Acid (Active Comparator): Topical application of 0.2% hyaluronic acid gel will be placed immediately in palatal donor site after free gingival graft harvesting and covered by periodontal pack
  Interventions: Drug: Topical application of 0.2% hyaluronic acid gel
- Platelet Rich Fibrin (Experimental): Palatal donor site will receive a platelet rich fibrin and then will be sutured by criss cross suture then covered by periodontal pack.
  Interventions: Biological: Platelet rich fibrin

INTERVENTIONS:
Drug: Topical application of 0.2% hyaluronic acid gel — Topical application of 0.2% hyaluronic acid gel will be placed immediately in palatal donor site after free gingival graft harvesting
  Other Names: gengigel
  Arms: Topical application 0.2%Hyaluronic Acid
Biological: Platelet rich fibrin — Placement of Platelet rich fibrin in the palatal donor sie after free gingival graft harvesting and suturing by criss cross sutured then covered by periodontal pack.
  Arms: Platelet Rich Fibrin

SUMMARY:
Comparative study to assess the efficacy of topical application of 0.2% hyaluronic acid vs platelet rich fibrin in decreasing a postoperative pain following free gingival graft procedure .

.

DETAILED DESCRIPTION:
- Patients of both groups will be subjected to:

1. Case history including personal data, medical, surgical history and family history.
2. Clinical Examination.

After local infiltration of anesthesia, an adequate size of supraperiosteal recipient bed was prepared to receive the palatal graft of 15 mm mesio-distal width with 8 mm apico-coronal extension.. The free gingival graft extended from the mesial line angle upper 5 and distal line angle of upper 6 .

The coronal horizontal incision, will be 15 mm long, at least 2 mm apical from the gingival margin. A second horizontal incision will be drawn 8 mm apico coronal . Care will be taken to obtain a graft thickness of 1.5 mm. Thickness will be measured at the central point of the graft during the surgery by using an endodontic file then the grafts will be positioned, and firmly adapted to the bed, and stabilized with simple periosteal sutures.

Preparation of platelet rich fibrin:( intervention group) The classic PRF protocol was introduced by Choukroun & coworkers. PRF requires around 10 ml of blood to be collected from the forearm of patient without anticoagulant in a glass coated plastic tubes. After collection, the blood will be quickly subjected to centrifugation at 2700-3000 rpm for 12 minutes. After the completion of cycle, the blood become separated into three distinct layers; platelet poor plasma at the top, PRF in the middle and a red blood corpuscular base in the bottom. Pliers will be inserted into the tube to gently grab the fibrin clot with attached RBC's. The clot thus obtained will be compressed to form plugs to be placed in the palatal donor site and stabilized by criss cross resorbable suture then covered by periodontal pack

control group Control group: As the intervention group but the palatal wound will receive a .2% hyaluronic acid gel then covered by periodontal dressing

..

ELIGIBILITY:
Inclusion Criteria for participants:

* Patients with mucogingival defects scheduled for free gingival graft
* Age at least 18 years.
* Not having any systemic disease that could compromise wound healing
* No previous periodontal surgery on the experimental sites.

Exclusion Criteria for participants:

* Systemic diseases that may be a contraindication for any surgeries.
* Loss of maxillary premolars and molars.
* Pregnancy or lactation
* Smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
post operative pain | 1 week
  Questionnaire will be used to evaluate the postoperative pain using visual analogue scale ( VAS) Min score Zero , Max score ten where zero is the best while ten is the worst

SECONDARY OUTCOMES:
wound healing | 2 months
  Early Wound Healing Index (EHI) , measuring unit Binary (YES/NO)

CONTACTS AND LOCATIONS:
Overall Officials: Mona M Shoeib, P.H.D, Study Director — Cairo University
Locations (1):
- Faculty of Dental Medicine - Cairo University -, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No